CLINICAL TRIAL: NCT00217295
Title: A Safety Study of Combination Treatment With Avonex and Placebo-Controlled Dosing of Topamax in Relapsing-Remitting Multiple Sclerosis.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Multiple Sclerosis Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MSI-101; BiogenIdec; Ortho-McNeil
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2005-09-22 (Estimated); Status verified 2005-06

CONDITIONS: Multiple Sclerosis
Keywords: Relapsing-remitting multiple sclerosis; Brain atrophy; Disease progression
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting; Disease Progression | interventions — Interferon beta-1a; Topiramate

INTERVENTIONS:
Drug: Avonex and Topamax

SUMMARY:
This is a clinical trial in relapsing-remitting Multiple Sclerosis to determine if Topamax added to Avonex has a neuroprotective effect as measured by the brain parenchymal fraction ( a measure of brain shrinkage) and by clinical assessment scores to evaluate disease progression.

DETAILED DESCRIPTION:
The protocol requires all participants to be treated with Avonex and in addition patients will be blindly assigned to either a group who receive Topamax or a placebo control. Repeated neurological and clinical examinations are performed with laboratory tests to determine any possible adverse drug effects. The scaled neurologic examinations (EDSS and MSFC) and brain MRI's are done at regular intervals to evaluate possible treatment effects.

ELIGIBILITY:
Inclusion Criteria:

Relapsing-remitting multiple sclerosis

-

Exclusion Criteria:

Secondary progressive multiple sclerosis Contraindication to MRI Systemic disease Pregnancy -

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30
Dates: Start 2004-04; Study Completion 2007-12

PRIMARY OUTCOMES:
Safety and tolerability

SECONDARY OUTCOMES:
Brain atrophy on nMRI
Disease progression on EDSS and MSFC
Relapse rate

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey I Greenstein, MD, Principal Investigator — MSI
Locations (1):
- Multiple Sclerosis Institute, Philadelphia, Pennsylvania, United States